CLINICAL TRIAL: NCT00123071
Title: Variability of Ventricular Mass, Volume, and Ejection Fraction in Pediatric Cardiomyopathy Patients (A Study Conducted by the Pediatric Heart Network)
Brief Title: Variability of Ventricular Mass, Volume, & Ejection Fraction in Pediatric Cardiomyopathy Patients-Pediatric Heart Network
Acronym: VVV
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Sponsor
Other Study IDs: 236; U01HL068292 (NIH); U01HL068290 (NIH); U01HL068288 (NIH); U01HL068285 (NIH); U01HL068281 (NIH); U01HL068279 (NIH); U01HL068270 (NIH); U42 HL068269
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational study will provide data (variations in ventricular size and function) that are essential to designing and conducting clinical trials. In addition, the study will evaluate intra- and inter-study variability seen in echocardiography.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiomyopathy is an important cause of chronic disability and death in pediatric patients and currently accounts for approximately 50% of cardiac transplants performed during childhood. Left ventricular (LV) size and function are important independent predictors of outcome, and echocardiography is the primary way to assess ventricular function in children. Although there is extensive experience with this technology, data are limited on how ventricular function changes over time in children, which is a major impediment to conducting controlled trials of therapy in children.

This study has been approved by the Institutional Review Boards/Research Ethics Boards of all participating clinical centers:

Hospital for Sick Children, Toronto, Canada

Children's Hospital Boston, Boston, MA

Columbia College of Physicians and Surgeons, New York, NY

Children's Hospital of Philadelphia, Philadelphia, PA

Duke University Medical Center, Durham, NC

Brody School of Medicine at East Carolina University, Greenville, NC

Wake Forest Baptist Medical Center, Winston Salem, NC

Medical University of South Carolina, Charleston, SC

Primary Children's Medical Center, Salt Lake City, UT

Washington University, St. Louis, MO

DESIGN NARRATIVE:

This observational study will prospectively evaluate pediatric patients with dilated cardiomyopathy who are undergoing clinically indicated echocardiographic evaluation of LV function. Patients who undergo at least two echocardiograms 3 to 18 months apart will have their studies performed by the same ultrasonographer. All studies will be sent to the core laboratory for evaluation of variability in LV mass, volume, and ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Less than 22 years of age
* Any race
* Diagnosis of dilated cardiomyopathy
* LV and diastolic diameter greater than 5.5 cm (or z-score for BSA greater than 2) on the primary image acquisition from the first study echocardiogram
* LV ejection fraction less than 50% (or z-score for age less than -2) or shortening fraction less than 28% (or z-score for age less than -2) as measured on the primary image acquisition from the first study echocardiogram
* Disease onset greater than 2 months prior to screening
* Anticipated to undergo repeat evaluation at the same institution at least 3 months but not more than 13 months later
* Informed consent of parent(s) or legal guardian and assent of subject if required

Exclusion Criteria:

* Hypertrophic cardiomyopathy
* Restrictive cardiomyopathy
* Myocardial noncompaction (LV hypertrabeculation); patient is eligible for the study as long as the echocardiogram performed at the time of screening has no evidence of myocardial noncompaction
* Ventricular paced rhythm
* Atrial or ventricular ectopy at ratio greater than 1:4
* Suspected acute myocarditis
* Tachycardia-induced cardiomyopathy
* Congenital heart disease (repaired or unrepaired)
* Currently on intravenous inotropic support
* Current left ventricular assist device (LVAD) or extracorporeal membrane oxygenation (ECMO)
* Heart transplant waiting list status of 1A or 1B
* Co-morbid condition that precludes the ability to successfully obtain an echocardiogram according to the specifications of the study protocol

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients up to 22 years of age with dilated cardiomyopathy followed at participating clinical centers or newly diagnosed during the recruitment period
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Inter-study variability of echo measurements; variance at a single point in time and variance of change in measurements over time | Measured for up to 18 months

SECONDARY OUTCOMES:
Relative magnitude of the various sources of variability in echocardiographic outcomes in order to optimize operational procedures that can minimize variance | Measured for up to 18 months
Interstudy variability of echocardiographically-derived indices of LV systolic and diastolic function derived from m-mode, spectral Doppler, and tissue Doppler techniques used in pediatric patients with dilated cardiomyopathy | Measured for up to 18 months
Relationship of clinical status, including treatment, to the interstudy variability and repeatability of echocardiographic measurements. | Measured for up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sleeper, ScD, Principal Investigator — Carelon Research
Locations (8):
- United States (7):
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Selamet Tierney ES, Hollenbeck-Pringle D, Lee CK, Altmann K, Dunbar-Masterson C, Golding F, Lu M, Miller SG, Molina K, Natarajan S, Taylor CL, Trachtenberg F, Colan SD; Pediatric Heart Network Investigators. Reproducibility of Left Ventricular Dimension Versus Area Versus Volume Measurements in Pediatric Patients With Dilated Cardiomyopathy. Circ Cardiovasc Imaging. 2017 Nov;10(11):e006007. doi: 10.1161/CIRCIMAGING.116.006007. PMID 29133477
- [Derived] Lee CK, Margossian R, Sleeper LA, Canter CE, Chen S, Tani LY, Shirali G, Szwast A, Tierney ES, Campbell MJ, Golding F, Wang Y, Altmann K, Colan SD; Pediatric Heart Network Investigators. Variability of M-mode versus two-dimensional echocardiography measurements in children with dilated cardiomyopathy. Pediatr Cardiol. 2014 Apr;35(4):658-67. doi: 10.1007/s00246-013-0835-9. Epub 2013 Nov 22. PMID 24265000
- [Derived] Molina KM, Shrader P, Colan SD, Mital S, Margossian R, Sleeper LA, Shirali G, Barker P, Canter CE, Altmann K, Radojewski E, Tierney ES, Rychik J, Tani LY; Pediatric Heart Network Investigators. Predictors of disease progression in pediatric dilated cardiomyopathy. Circ Heart Fail. 2013 Nov;6(6):1214-22. doi: 10.1161/CIRCHEARTFAILURE.113.000125. Epub 2013 Oct 16. PMID 24132734
- [Derived] Colan SD, Shirali G, Margossian R, Gallagher D, Altmann K, Canter C, Chen S, Golding F, Radojewski E, Camitta M, Carboni M, Rychik J, Stylianou M, Tani LY, Selamet Tierney ES, Wang Y, Sleeper LA; Pediatric Heart Network Investigators. The ventricular volume variability study of the Pediatric Heart Network: study design and impact of beat averaging and variable type on the reproducibility of echocardiographic measurements in children with chronic dilated cardiomyopathy. J Am Soc Echocardiogr. 2012 Aug;25(8):842-854.e6. doi: 10.1016/j.echo.2012.05.004. Epub 2012 Jun 5. PMID 22677278